CLINICAL TRIAL: NCT04280692
Title: Safety and Feasibility of a Malaria Transmission Model in Semi-immune Kenyan Adults Using Plasmodium Falciparum Sporozoites
Brief Title: Controlled Human Malaria Infection Transmission Model - Phase A
Acronym: CHMI-TransMod
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely due to US FDA clinical hold on PfSPZ Challenge
Sponsor: University of Oxford (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other); Sanaria Inc. (Industry); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: KEMRI/SERU/CGMR-C/117/3759; OxTREC 48-18 (Other: Oxford Tropica Research Ethics Committee)
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Malaria,Falciparum
Keywords: PfSPZ; Kenya; Gametocytes; Transmission; CHMI; Challenge; semi-immune adults
MeSH Terms: conditions — Malaria, Falciparum | interventions — fanasil, pyrimethamine drug combination; piperaquine; Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: PfSPZ 6,400 (Experimental): Group 1 will receive a malaria infection by direct venous inoculation (DVI) with PfSPZ Challenge at a dose of 6,400 sporozoites.
  Group 1 will be randomised (1:1) to receive either sub-curative Sulfadoxine-Pyrimethamine (SP) (500mg/25mg) or Piperaquine (PIP) (480mg).
  Group 1 will receive a final curative treatment of Artemether-Lumefantrine (AL) with single low dose Primaquine (SLDPQ)
  Interventions: Biological: PfSPZ Challenge; Drug: Sulfadoxine-Pyrimethamine; Drug: Piperaquine; Drug: Artemether lumefantrine; Drug: Primaquine
- Group 1: PfSPZ 12,800 (Experimental): Group 2 will receive a malaria infection by direct venous inoculation (DVI) with PfSPZ Challenge at a dose of 12,800 sporozoites
  Group 2 will be randomised (1:1) to receive either sub-curative Sulfadoxine-Pyrimethamine (SP) (500mg/25mg) or Piperaquine (PIP) (480mg).
  Group 2 will receive a final curative treatment of Artemether-Lumefantrine (AL) with single low dose Primaquine (SLDPQ)
  Interventions: Biological: PfSPZ Challenge; Drug: Sulfadoxine-Pyrimethamine; Drug: Piperaquine; Drug: Artemether lumefantrine; Drug: Primaquine
- Group 3: PfSPZ 25,600 (Experimental): Group 3 will receive a malaria infection by direct venous inoculation (DVI) with PfSPZ Challenge at a dose of 25,600 sporozoites
  Group 3 will be randomised (1:1) to receive either sub-curative Sulfadoxine-Pyrimethamine (SP) (500mg/25mg) or Piperaquine (PIP) (480mg).
  Group 3 will receive a final curative treatment of Artemether-Lumefantrine (AL) with single low dose Primaquine (SLDPQ)
  Interventions: Biological: PfSPZ Challenge; Drug: Sulfadoxine-Pyrimethamine; Drug: Piperaquine; Drug: Artemether lumefantrine; Drug: Primaquine

INTERVENTIONS:
Biological: PfSPZ Challenge — Aseptic, purified, cryopreserved Plasmodium falciparum sporozoites
  Other Names: NF54 Plasmodium falciparum malaria challenge
Drug: Sulfadoxine-Pyrimethamine — Sub-curative 500mg/25mg single dose regimen
  Other Names: Fansidar
Drug: Piperaquine — Sub-curative 480mg single dose regimen
  Other Names: Piperaquine Phosphate
Drug: Artemether lumefantrine — Three day curative regimen 20mg/120mg
  Other Names: Coartem
Drug: Primaquine — Single low dose regimen 0.25 mg base/kg

SUMMARY:
This is to develop a model to test the efficacy of vaccines and/or drugs designed to block transmission of malaria to mosquitoes and to identify the targets of transmission-blocking immunity to malaria.

DETAILED DESCRIPTION:
Malaria is a disease of major public health importance. The only vaccine available is partially effective and targets the pre-erythrocytic stages of the life cycle. Thus, there is a need to identify other potential vaccine targets as well as to develop models to test vaccine efficacy, especially that of transmission-blocking vaccines. Controlled human malaria infection (CHMI) has been shown to be an important tool for the assessment of the efficacy of novel malaria vaccines and drugs. CHMI also allows for the evaluation of immunity to malaria and monitoring of parasite growth rates in vivo. This is particularly useful in individuals from endemic areas with varying levels of exposure and immunity to malaria. Thus, CHMI in individuals with prior exposure to malaria has potential to accelerate malaria vaccine development. In this study, the aim is to use CHMI in semi-immune adults to develop a model to assess transmissibility of malaria infection to mosquitoes, to study immune responses that are directed against sexual stages that might block transmission, and as a platform to test vaccines. To achieve this, the study will be carried out in two phases A (N=45 participants) and B (N=60 participants) over a period of 4-6months. Parasite dose will be varied in individuals enrolled for CHMI and use of low-doses of anti-malarial drugs to promote the production of gametocytes in vivo (Phase A) and demonstrate transmissibility in mosquito feeding assays (Phase B). Thus, the main outcomes of the study will be: (1) optimisation of sporozoite dose for infections success in individuals with moderate-high malaria exposure; (2) use of sub-curative anti-malaria treatment for induction of gametocytes; and (3) infection of mosquitoes in mosquito feeding assays by induced gametocytes. To achieve this, up to 250 semi-immune adults will be recruited from known areas of malaria endemicity in Kenya with varying exposure to malaria undergo screening procedures after informed consent to enrol 105 individuals to conduct CHMI studies with serial quantitative polymerase chain reaction (PCR) to measure asexual parasite growth and induction of transmission stages in vivo. In addition, comprehensively characterize immunity and identify targets in relation to function assessed by various laboratory assays.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 to 45 years.
2. Able and willing (in the Investigator's opinion) to comply with all study requirements.
3. Informed consent.
4. Use of effective method of contraception for duration of study (women only). We will ask the female volunteers to come with their family planning records to verify. Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly, in accordance with the product label. Examples of these include: combined oral contraceptives; injectable progestogen; implants of etenogestrel or levonorgestrel; intrauterine device or intrauterine system; male partner sterilisation at least 6 months prior to the female subject's entry into the study, and the relationship is monogamous; male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository); and male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).

Exclusion Criteria:

1. Body weight of less than 50kg or body mass index (BMI) less than 18 or greater than 25 kg/m2 at screening.
2. Use of systemic antibiotics with known antimalarial activity within 30 days of administration of PfSPZ Challenge (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
3. Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
4. Current participation in another clinical trial or recent participation within 12 weeks of enrolment.
5. Prior receipt of an investigational malaria vaccine.
6. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed). This will also include Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) positivity.
7. Use of immunoglobulins or blood products within 3 months prior to enrolment.
8. Any serious medical condition reported or identified during screening that increases the risk of CHMI.
9. Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
10. Women only; pregnancy, or an intention to become pregnant during the duration of the study.
11. Sickle cell trait or disease.
12. History of drug or alcohol abuse.
13. Known hypersensitivity to or contraindications for use of artemether-lumefantrine, chloroquine, piperaquine, primaquine, sulfadoxine-pyrimethamine, or history of severe (allergic) reactions to mosquito bites.
14. Confirmed gametocyte positivity at screening and/or a day before challenge
15. Confirmed parasite positive by PCR a day before challenge i.e. at C-1. Exclusion Criterion on Day of Challenge

    * Acute disease, defined as moderate or severe illness with or without fever (temperature >37.5 degrees Celcius).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety and optimisation of sporozoite dose for infections success in individuals with moderate-high malaria exposure | Up to 42 days post infection with PfSPZ challenge
  Magnitude and frequency of adverse events in the study groups
Prevalence of gametocytes | Up to 42 days post infection with PfSPZ challenge
  Prevalence of gametocytes as determined by qRT-PCR

SECONDARY OUTCOMES:
Use of sub-curative anti-malaria treatment for induction of gametocytes | Up to 42 days post infection with PfSPZ challenge
  Density of gametocytes as measured by qRT-PCR
Peak density and time point of gametocytaemia | Up to 42 days post infection with PfSPZ challenge
  Peak density and peak time point of gametocytes by drug-regimen and determine the area under the curve of density over time

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI-Wellcome Trust Research Programme, Kilifi, Kenya